CLINICAL TRIAL: NCT04492384
Title: Analysis of Chronic Non-infectious Diseases Dynamics After COVID-19 Infection in Adult Patients
Acronym: ACTIV
Status: Completed | Type: Observational
Sponsor: Eurasian Association of Therapists (Other)
Responsible Party: Principal Investigator, Tamara Kriukova, Head of Organizational Committee, Eurasian Association of Therapists
Other Study IDs: ACTIV11062020
Record Dates: First submitted 2020-07-27; First posted 2020-07-30 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Covid19; SARS-CoV-2 Infection; Pneumonia; Copd; CKD; Cardiac Event; Overweight and Obesity; Cardiovascular Diseases; Diabetes; Hypertension; Coronary Heart Disease
MeSH Terms: conditions — COVID-19; Pneumonia; Pulmonary Disease, Chronic Obstructive; Cardiovascular Diseases; Overweight; Obesity; Diabetes Mellitus; Hypertension; Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- inpatients: Patients treated from COVID-19 in hospital
  Interventions: Other: non-interventional
- outpatients: Patients treated from COVID-19 at home
  Interventions: Other: non-interventional

INTERVENTIONS:
Other: non-interventional — Interview on health conditions

SUMMARY:
Non-commercial depersonalized multi-centered registry study on analysis of chronic non-infectious diseases dynamics after SARS-CoV-2 infection in adults.

DETAILED DESCRIPTION:
Non-commercial depersonalized multi-centered registry study on analysis of chronic non-infectious diseases dynamics after SARS-CoV-2 infection in cohort of Russian adult patients.

Retrospective analysis of medical histories and outcomes in adults with pre-existing conditions after SARS-CoV-2 infection and prospective monitoring of health status during 3, 6 and 12 months after discharge. Comorbidities worsening risk factors measuring through evaluation of range of indicators such as dynamics of diabetes, CKD, COPD, bronchial astma, incidence of hypertonic crises, vascular events and others.

ELIGIBILITY:
Inclusion Criteria:

* Suspected or confirmed COVID-19.

Exclusion Criteria:

* Refuse to be involved in study;
* Age under 18 years.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Anonymized male and female patients over 18 years infected COVID-19 recieved inpatient or outpatient care
Sampling Method: Probability Sample
Enrollment: 6396 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2020-11-29 (Actual); Study Completion 2021-11-29 (Actual)

PRIMARY OUTCOMES:
rate of non-infectious diseases | 12 month since a moment of request of medical help
  percentage of patients with non-infectious diseases relating to overall number of patients registered in study
severity of COVID-19 depending on pre-existing diseases | 12 month since a moment of request of medical help
  correlation between number of patients with COVID-19 of various severity and number of pre-existing conditions and their severity among these groups
disability registration / change of disability status | 12 month since a moment of request of medical help
  Registration of disability or change of disability status
rate of letal outcomes | 12 month since a moment of request of medical help
  rate of deaths among registered participants
rate of letal outcomes depending on pre-existing disease | 12 month since a moment of request of medical help
  correlation between number of deaths and pre-existing diseases

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Arutyunov, professor, Study Chair — Eurasian Association of Therapists
Locations (1):
- Eurasian Association of Therapists, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shchepikhin EI, Shmelev EI, Ergeshov AE. [Pulmonary fibrosis after a new coronavirus infection - versions and controversies: A review]. Ter Arkh. 2024 Apr 16;96(3):298-302. doi: 10.26442/00403660.2024.03.202632. Russian. PMID 38713047
- [Derived] Arutyunov GP, Tarlovskaya EI, Arutyunov AG, Belenkov YN, Konradi AO, Lopatin YM, Rebrov AP, Tereshchenko SN, Chesnikova AI, Hayrapetyan HG, Babin AP, Bakulin IG, Bakulina NV, Balykova LA, Blagonravova AS, Boldina MV, Vaisberg AR, Galyavich AS, Gomonova VV, Grigorieva NY, Gubareva IV, Demko IV, Evzerikhina AV, Zharkov AV, Kamilova UK, Kim ZF, Kuznetsova TY, Lareva NV, Makarova EV, Malchikova SV, Nedogoda SV, Petrova MM, Pochinka IG, Protasov KV, Protsenko DN, Ruzanau DY, Sayganov SA, Sarybaev AS, Selezneva NM, Sugraliev AB, Fomin IV, Khlynova OV, Chizhova OY, Shaposhnik II, Sh'ukarev DA, Abdrahmanova capital A, CyrillicK, Avetisian SA, Avoyan HG, Azarian KK, Aimakhanova GT, Ayipova DA, Akunov AC, Alieva MK, Aparkina AV, Aruslanova OR, Ashina EY, Badina OY, Barisheva OY, Batchayeva AS, Bitieva AM, Bikhteyev IU, Borodulina NA, Bragin MV, Budu AM, Bykova GM, Vagapova KR, Varlamova DD, Vezikova NN, Verbitskaya EA, Vilkova OE, Vinnikova EA, Vustina VV, Galova EA, Genkel VV, Gorshenina EI, Gostishev RV, Grigorieva EV, Gubareva EY, Dabylova GM, Demchenko AI, Dolgikh OY, Duyshobayev MY, Evdokimov DS, Egorova KE, Ermilova AN, Zheldybayeva AE, Zarechnova NV, Zimina YD, Ivanova SY, Ivanchenko EY, Ilina MV, Kazakovtseva MV, Kazymova EV, Kalinina YS, Kamardina NA, Karachenova AM, Karetnikov IA, Karoli NA, Karsiev MK, capital KA, Cyrillicaskaeva DS, Kasymova KF, Kerimbekova ZB, Kerimova AS, Kim ES, Kiseleva NV, Klimenko DA, Klimova AV, Kovalishena OV, Kolmakova EV, Kolchinskaya TP, Kolyadich MI, Kondriakova OV, Konoval MP, Konstantinov DY, Konstantinova EA, Kordukova VA, Koroleva EV, Kraposhina AY, Kriukova TV, Kuznetsova AS, Kuzmina TY, Kuzmichev KV, Kulchoroevna CK, Kuprina TV, Kouranova IM, Kurenkova LV, Kurchugina NY, Kushubakova NA, Levankova VI, Lyubavina NA, Magdeyeva NA, Mazalov KV, Majseenko VI, Makarova AS, Maripov AM, Marusina AA, Melnikov ES, Moiseenko NB, Muradova FN, Muradyan RG, Musaelian SN, Myshak AO, Nekaeva ES, Nikitina NM, Ogurlieva BB, Odegova AA, Omarova YV, Omurzakova NA, Ospanova SO, Pahomova EV, Petrov LD, Plastinina SS, Pogrebetskaya VA, Polyakov DS, Ponomarenko EV, Popova LL, Prokofeva NA, Pudova IA, Rakov NA, Rahimov AN, Rozanova NA, Serikbolkyzy S, Simonov AA, Skachkova VV, Soloveva DV, Soloveva IA, Subbotin AK, Sukhomlinova IM, Sushilova AG, Tagayeva DR, Titojkina YV, Tikhonova EP, Tokmin DS, Tolmacheva AA, Torgunakova MS, Trenogina KV, Trostianetckaia NA, Trofimov DA, Tulichev AA, Tursunova AT, Ulanova ND, Fatenkov OV, Fedorishina OV, Fil TS, Fomina IY, Fominova IS, Frolova IA, Tsvinger SM, Tsoma VV, Cholponbaeva MB, Chudinovskikh TI, Shevchenko OA, Sheshina TV, Shishkina EA, Shishkov KY, Sherbakov SY, Yausheva EA. [ACTIV SARS-CoV-2 registry (Analysis of Chronic Non-infectious Diseases Dynamics After COVID-19 Infection in Adult Patients). Assessment of impact of combined original comorbid diseases in patients with COVID-19 on the prognosis]. Ter Arkh. 2022 Jan 15;94(1):32-47. doi: 10.26442/00403660.2022.01.201320. Russian. PMID 36286918
- [Derived] Tarlovskaya EI, Arutyunov AG, Konradi AO, Lopatin YM, Rebrov AP, Tereshchenko SN, Chesnikova AI, Hayrapetyan HG, Babin AP, Bakulin IG, Bakulina NV, Balykova LA, Blagonravova AS, Boldina MV, Vaisberg AR, Galyavich AS, Gomonova VV, Grigorieva NY, Gubareva IV, Demko IV, Evzerikhina AV, Zharkov AV, Kamilova UK, Kim ZF, Kuznetsova TY, Lareva NV, Makarova EV, Malchikova SV, Nedogoda SV, Petrova MM, Pochinka IG, Protasov KV, Protsenko DN, Ruzanau DY, Sayganov SA, Sarybaev AS, Selezneva NM, Sugraliev AB, Fomin IV, Khlynova OV, Chizhova OY, Shaposhnik II, Shsmall es, Cyrillicukarev DA, Abdrahmanova AK, Avetisian SA, Avoyan HG, Azarian KK, Aimakhanova GT, Ayipova DA, Akunov AC, Alieva MK, Aparkina AV, Aruslanova OR, Ashina EY, Badina OY, Barisheva OY, Batchayeva AS, Bitieva AM, Bikhteyev IU, Borodulina NA, Bragin MV, Budu AM, Burygina LA, Bykova GA, Vagapova KR, Varlamova DD, Vezikova NN, Verbitskaya EA, Vilkova OE, Vinnikova EA, Vustina VV, Gsmall a, Cyrilliclova EA, Genkel VV, Gorshenina EI, Gostishev RV, Grigorieva EV, Gubareva EY, Dabylova GM, Demchenko AI, Dolgikh OY, Duyshobayev MY, Evdokimov DS, Egorova KE, Ermilova AN, Zheldybayeva AE, Zarechnova NV, Zimina YD, Ivanova SY, Ivanchenko EY, Ilina MV, Kazakovtseva MV, Kazymova EV, Kalinina YS, Kamardina NA, Karachenova AM, Karetnikov IA, Karoli NA, Karpov OV, Karsiev MK, capital KA, Cyrillicaskaeva DS, Kasymova KF, Kerimbekova ZB, Kerimova AS, Kim ES, Kiseleva NV, Klimenko DA, Klimova AV, Kovalishena OV, Kolmakova EV, Kolchinskaya TP, Kolyadich MI, Kondriakova OV, Konoval MP, Konstantinov DY, Konstantinova EA, Kordukova VA, Koroleva EV, Kraposhina AY, Kriukova TV, Kuznetsova AS, Kuzmina TY, Kuzmichev KV, Kulchoroeva CK, Kuprina TV, Kouranova IM, Kurenkova LV, Kurchugina NY, Kushubakova NA, Levankova VI, Levin Mcapital IE, Cyrillic, Lyubavina NA, Magdeyeva NA, Mazalov KV, Majseenko VI, Makarova AS, Maripov AM, Marusina AA, Melnikov ES, Moiseenko NB, Muradova FN, Muradyan RG, Myshak AO, Nikitina NM, Ogurlieva BB, Odegova AA, Omarova YM, Omurzakova NA, Ospanova SO, Pahomova EV, Petrov LD, Plastinina SS, Pogrebetskaya VA, Polyakov DS, Ponomarenko EV, Popova LL, Prokofeva NA, Pudova IA, Rakov NA, Rakhimov AN, Rozanova NA, Serikbolkyzy S, Simonov AA, Skachkova VV, Soloveva DV, Soloveva IA, Sokhova FM, Subbotin AK, Sukhomlinova IM, Sushilova AG, Tagayeva DR, Titojkina YV, Tikhonova EP, Tokmin DS, Tolmacheva AA, Torgunakova MS, Trenogina KV, Trostianetckaia NA, Trofimov DA, Tulichev AA, Tursunova AT, Ulanova ND, Fatenkov OV, Fedorishina OV, Fil TS, Fomina IY, Fominova IS, Frolova IA, Tsvinger SM, Tsoma VV, Cholponbaeva MB, Chudinovskikh TI, Shevchenko OA, Sheshina TV, Shishkina EA, Shishkov KY, Sherbakov SY, Yausheva EA, Musaelian SN, Belenkov YN, Arutyunov GP. Analysis of influence of background therapy for comorbidities in the period before infection on the risk of the lethal COVID outcome. Data from the international ACTIV SARS-CoV-2 registry (<<Analysis of chronic non-infectious diseases dynamics after COVID-19 infection in adult patients SARS-CoV-2>>). Kardiologiia. 2021 Sep 30;61(9):20-32. doi: 10.18087/cardio.2021.9.n1680. English, Russian. PMID 34713782
- See also: results of the first interim statistical analysis (1000 patients) — https://russjcardiol.elpub.ru/jour/article/view/4165
- See also: study design — https://lib.ossn.ru/jour/article/view/1519
- See also: design of observatinal studies "Analysis of Chronic Non-infectious Diseases Dynamics After COVID-19 Infection in Adult Patients" and "Analysis of Health Status of Сomorbid Adult COVID-19 Patients Hospitalised in Second Wave of SARS-CoV-2 Infection" — http://russjcardiol.elpub.ru/jour/article/view/4358/
- See also: Analysis of predictors of short-term adverse outcomes in COVID-19. Data from the international ACTIV SARS-CoV-2 registry — http://russjcardiol.elpub.ru/jour/article/view/4470?locale=ru_RU
- See also: Analysis of influence of background therapy for comorbidities in the period before infection on the risk of the lethal COVID outcome. Data from the international ACTIV SARS-CoV-2 registry — http://lib.ossn.ru/jour/article/view/1680
- See also: Clinical features of post-COVID period. Results of an international registry "ACTIV SARS-CoV-2". Preliminary data. (6 month follow-up) — http://russjcardiol.elpub.ru/jour/article/view/4708
- See also: Assessment of impact of combined original comorbid diseases in patients with COVID-19 on the prognosis — https://ter-arkhiv.ru/0040-3660/article/view/71639
- See also: Comparative analysis of echocardiographic and electrocardiographic data of survivors and deceased patients with COVID-19 (sub-analysis of the international register "Dynamics analysis of comorbidities in SARS-CoV-2 survivors") — https://russjcardiol.elpub.ru/jour/article/view/4855
- See also: Lipid profile in hospitalized patients with COVID-19 depending on the outcome of its acute phase: data from the international registry "Dynamics analysis of comorbidities in SARS-CoV-2 infection survivors" — https://russjcardiol.elpub.ru/jour/article/view/5042
- See also: The impact of carbohydrate metabolism disorders on the early and long-term clinical outcomes of patients with COVID-19 according to the AKTIV and AKTIV 2 registries. — https://www.probl-endojournals.ru/jour/article/view/13175
- See also: Impact of Kidney Damage on the Course and Prognosis of COVID-19 Infection According to the International Registry "Analysis of Chronic Non-Infectious Diseases Dynamics After Covid-19 Infection in Adult Patients" — https://www.medarhive.ru/jour/issue/view/73/showToc
- See also: Impact of heart failure on all-cause mortality in COVID-19: findings from the Eurasian International Registry — https://pubmed.ncbi.nlm.nih.gov/36519220/